CLINICAL TRIAL: NCT01742793
Title: An Open Label, International, Multi-centre, Phase I/IIa Study of Lenalidomide (Revlimid) and Romidepsin (Istodax) for Relapsed /Refractory Hodgkin Lymphoma, Mature T-cell Lymphoma and Multiple Myeloma. (RId Study)
Acronym: RID
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to withdrawal of institutional support, Phase II never began.
Sponsor: Yale University (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Principal Investigator, Francine Foss, Principal Investigator, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1112009392; 115541 (Other: FDA)
Record Dates: First submitted 2012-11-21; First posted 2012-12-05 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2017-02

CONDITIONS: Hodgkin's Lymphoma; Mature T-cell Lymphoma; Multiple Myeloma
Keywords: relapsed /refractory Hodgkin lymphoma; mature T-cell lymphoma; multiple myeloma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell; Multiple Myeloma | interventions — Lenalidomide; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm L: subjects with lymphoma (Experimental): The following dosing steps will be applied to the dose-escalation, phase-I component of the study for patients with lymphoma who are eligible to enter Arm L:
  Dose Level Arm L Lenalidomide dose Oral Romidepsin Dose Intravenous
  * 2 10mg D1-7, D15-21 6mg D1, 8, 15
  * 1 10mg D1-7, D15-21 8mg D1, 8, 15
    1. 10mg D1-21 8mg D1, 8, 15 2 15mg D1-21 8mg D1, 8, 15 3 15mg D1-21 10mg D1, 8, 15 4 15mg D1-21 12mg D1, 8, 15 5 15mg D1-21 14mg D1, 8, 15 6 25mg D1-21 14mg D1, 8, 15
       * The first patient in arm L will be entered into the study at dosing level one.
  Interventions: Drug: lenalidomide (Revlimid) and romidepsin (Istodax)
- Arm M: subjects with myeloma (Experimental): The following dosing steps will be applied to the dose-escalation, phase-I component of the study for patients with myeloma who are eligible to enter Arm M:
  Dose Level Arm M Lenalidomide dose Oral Romidepsin Dose Intravenous Dexamethasone
  * 2 15mg D1-7, D15-21 6mg D1, 8, 15 20mg D1,8,15,22
  * 1 15mg D1-7, D15-21 8mg D1, D8, 15 20mg D1,8,15,22
    1. 15mg D1-21 8mg D1, 8, 15 20mg D1,8,15,22 2 25mg D1-21 8mg D1, 8, 15 20mg D1,8,15,22 3 25mg D1-21 10mg D1, 8, 15 20mg D1,8,15,22 4 25mg D1-21 12mg D1, 8, 15 20mg D1,8,15,22 5 25mg D1-21 14mg D1, 8, 15 20mg D1,8,15,22
       * The first patient in arm M will be entered into the study at dosing level one.
  Interventions: Drug: lenalidomide (Revlimid) and romidepsin (Istodax)

INTERVENTIONS:
Drug: lenalidomide (Revlimid) and romidepsin (Istodax)

SUMMARY:
The study hypothesis is that lenalidomide and romidepsin (and dexamethasone for patients with myeloma) will have an acceptable toxicity profile and that in combination will have sufficient activity in the target population (including those previously refractory to HDACi monotherapy) to warrant further investigation.

DETAILED DESCRIPTION:
Summary of rationale:

1. As individual agents, both the histone deacetylase inhibitors and lenalidomide have significant activity in each of the diseases in this study;
2. There is potential for the agents to synergize (to improve upon the response rates as there are both overlapping and disparate mechanisms of action.) Both agents may synergize to induce cell death through caspase 8-mediated and other mechanisms; both induce p21 and cell cycle arrest; both agents have anti-angiogenic effects; both are likely to interfere with PI3K/Akt signaling. One particularly attractive aspect of this combination is the potential for synergistic immunological effects, particularly related to T-cell polarization, NK cell activation, STAT signaling and cytokine production, as discussed above;
3. With respect to PTCL, CTCL and HL, there is a clear path for further drug development and registration if this trial proves that this is a safe and efficacious combination;
4. Myeloma is incurable and this is due to the persistence of a drug-resistant sub-clone of tumor-propagating cells that is drug insensitive. Preclinical data suggests that both HDACi and lenalidomide may target these tumor-propagating cells. This argues for examining this combination as part of early treatment in these diseases. This trial is the first step to examine the feasibility of combining an HDACi with what is front-line therapy in myeloma in the USA - lenalidomide.
5. Incorporating three separate arms (as opposed to three separate studies) will allow;

   i. The investigators to accumulate data on this novel combination across the three groups and evaluate the toxicity profiles to make informed decisions around dose-escalation. Because it is a single study, valid comparisons can be made across the groups, which would not be possible if they were separate studies.

   ii. combined and simplified collection of correlative tests across the three studies.

   This study was terminated and Phase 2 portion never was initiated.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a biopsy-proven diagnosis of one of the following malignancies that meets the additional disease-specific inclusion criteria.

   A. Mature T-Cell lymphoma. The following entities are eligible. PTCL or CTCL (including MF and SS) but excluding adult T-cell leukemia/lymphoma, primary cutaneous CD30+ lymphoma, lymphomatoid papulosis, and NK or LGL leukemia.(The complete WHO classification of T-cell lymphoma can be found in the appendices).
   1. Peripheral T-cell lymphoma: patients must have relapsed or progressed after: at least one prior chemotherapy-based treatment, or not suitable for a conventional chemotherapeutic approach as judged by the investigator.
   2. Sezary syndrome/ Mycosis Fungoides: patients must have relapsed or progressed after at least one prior systemic therapy.

   B. Hodgkin lymphoma
   1. At least one prior chemotherapy-based treatment.
   2. Prior autograft in those eligible for autologous transplantation according to institutional guidelines.

   C. Myeloma
   1. Relapsed after at least one prior systemic therapy that includes thalidomide (unless intolerant or contraindicated) or lenalidomide. Those who have received prior lenalidomide must have had a response that exceeded 6 months.
   2. Patients who are candidates for autologous stem cell transplant in first remission are not eligible.
   3. Patients must have failed/relapsed after bortezomib therapy.
2. ECOG performance status <2
3. Age >18 years.
4. Life expectancy ≥90 days.
5. Patients must have normal organ and marrow function as defined below:

   absolute neutrophil count >1.0 x109/L (or greater than 0.75x109/L if >50% plasma cells or >50% lymphoma in the bone marrow) Neutrophil count must not be supported by G-CSF prior to study entry. platelets >100 x109/L (or >75 x 109 if >50% plasma cells or >50% lymphoma in the bone marrow).

   (Transfusion to achieve these goals would not qualify the patient) total bilirubin <1.5x the institutional upper limit of normal. (<2.5x for Gilbert's disease).

   AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal

   Creatinine clearance >60 mL/min/1.73 m2 in the dose escalation phase, and >30 mL/min/1.73 m2 in phase II.

   Serum potassium & magnesium Serum potassium ≥3.8 mmol/L Serum magnesium ≥1.8mg/dL /0.75mmol/L (supplementation is allowed)
6. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

1. Patients receiving any other investigational agents within 4 weeks.
2. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not adequately recovered from grade III/IV adverse events due to agents administered more than 4 weeks earlier.
3. Prior exposure to lenalidomide, in patients with myeloma, except if a response (including stable disease) was maintained for at least 6 months. (Washout period of 4 weeks required)
4. Prior treatment with HDAC inhibitor (not including sodium valproate for neurological or psychiatric disorders), except if response (including stable disease) was maintained for at least 3 months. (Washout period of 4 weeks required)
5. Concomitant treatment with sodium valproate (washout 4 weeks required).
6. Central nervous system involvement by lymphoma or myeloma.
7. A history of allergic reaction to romidepsin or lenalidomide, boron or mannitol.
8. A history of Gr III/IV drug-related non-hematological toxicity, excluding thromboembolism or sepsis, in a prior exposure to either lenalidomide or a histone deacetylase inhibitor.
9. Concomitant corticosteroid except for patients on a stable dose of ≤10mg prednisone/day for at least 4 weeks prior to screening.
10. Congenital long QT syndrome, or a QTc interval >450 milliseconds
11. Patients who have had a myocardial infarction within twelve months of study entry.
12. Patients who have active coronary artery disease (for example NYHA class II or above angina).

    Any patient in whom coronary artery disease is suspected should be referred for a cardiology consultation and if active myocardial ischemia is demonstrated, the patient should be excluded. If a non-invasive imaging study is equivocal, it may be necessary to proceed to coronary angiography.
13. Patients with a baseline ECG showing evidence of cardiac ischaemia (ST depression of ≥2mm)
14. Patients with NYHA-class congestive heart failure ≥II
15. Patients with cardiac ejection fraction less than the institutional lower limited of normal by a gated heart-pool scan, or echocardiogram.
16. Patients with a history of sustained VT, VF, torsade de pointes or cardiac arrest unless that issue is currently managed with an implantable cardioverter defibrillator (AICD).
17. Patients with a cardiomyopathy of any cause.
18. Patients with uncontrolled hypertension ie. SBP ≥160mmHg or DBP ≥95mmHg
19. Patients with cardiac arrythmia requiring anti-arrythmic medication other than a beta blocker or calcium channel blocker. Patients in who digitalis can not be discontinued are excluded from the study.
20. Patients with mobitz-II second degree heart block that do not have a pacemaker.

    1. Patients with first degree or Mobitz-I second degree block, bradyarrhythmia or sick sinus syndrome require holter monitoring and evaluation for eligibility by a cardiologist.
    2. Patients with other cardiac disease may be excluded at the discretion of the PI following consultation with a cardiologist.
21. Patients who require concomitant use of drugs known to cause significant prolongation of the QT interval.
22. Patients who require concomitant use of warfarin, due to potential for drug interaction.
23. Pregnancy in female patients. Lactating females must agree not to breast feed while taking lenalidomide.
24. Patients with known HIV infection.
25. Patients with known Hepatitis B infection.
26. Prior allotransplantation, unless the patient has been completely weaned off immunosuppressive agents for ≥3 months.
27. Myeloma, patient who is a candidate for autologous stem cell transplant
28. Pre-existing motor or sensory neuropathy ≥ grade 3.
29. Other serious and / or uncontrolled medication condition
30. Prior diagnosis of cancer that was:

    1. more than 3 years prior to current diagnosis with estimated clinical expectation of progression greater than 10% within next 2 years.
    2. within 3 years of current diagnosis with the exception of successfully treated basal cell or squamous cell skin carcinoma, carcinoma in situ of the cervix or localised cancer treated curatively with local therapy only.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Overall Rate of Clinical Response (Complete Response + Partial Response) | 12 months
  Overall response rate is a combination of partial response and complete response according to specific response criteria that will be used throughout the study.
Overall Rate of Clinical Response (Complete Response + Partial Response) | 24 months
  Overall response rate is a combination of partial response and complete response according to specific response criteria that will be used throughout the study.

SECONDARY OUTCOMES:
Rate of Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 70 months.

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

REFERENCES:
- See also: Yale Cancer Center Website — http://www.yalestudies.org